CLINICAL TRIAL: NCT06231277
Title: Phase I Clinical Trial of Safety, Tolerability and Pharmacokinetics of BH002 in Patients With Advanced Solid Tumors
Brief Title: Phase I Clinical Trial of BH002 in Patients With Advanced Solid Tumors
Acronym: BH002-Ⅰ-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhuhai Beihai Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH002-Ⅰ-101; CTR20220209 (Other: NMPA)
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumours
Keywords: Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BH002 (Experimental): Every 21 days constitutes a treatment cycle, and administration begins on the first day of each cycle
  Interventions: Drug: BH002

INTERVENTIONS:
Drug: BH002 — Every 21 days constitutes a treatment cycle, and administration begins on the first day of each cycle

SUMMARY:
The goal of this clinical trial is to about in Patients With Advanced Solid Tumors. The main question[s] it aims to answer are:

* question 1:Evaluating the tolerability of BH002 injection in Chinese patients with advanced solid tumors
* question 2:Obtain the pharmacokinetic (PK) characteristics of BH002 injection in Chinese patients with advanced solid tumors

DETAILED DESCRIPTION:
Subjects will be administered BH002 intravenously. It is expected that there will be 2 to 4 dose groups, with 3 to 6 subjects enrolled in each group. The doses from low to high are 15 mg/m2,20 mg/m2,25 mg/m2,30 mg/m2,35 mg/m2. Subjects were injected with BH002 intravenously on the first day of each cycle, once during a 3-week period.

The dose escalation for this trial will be 20mg/m2 as the starting dose. According to the traditional "3+3" dose escalation principle, 3 subjects are planned to be enrolled in each dose group at the same time. Safety, tolerability, and dose-limiting toxicities (DLTs) will be assessed within 21 days of first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female.
2. Patients were diagnosed advanced solid tumors by histology or cytology (preferably prostate cancer, gastric cancer, non-small cell lung cancer, breast cancer, esophageal cancer, head and neck squamous cell carcinoma, ovarian cancer, liposarcoma, etc.) whose disease progresses after standard treatment.
3. ECOG score 0~2, expected survival time ≥3 months.
4. Have adequate hematology and organ function, and meet the following conditions based on laboratory test results within 7 days before the first dose:1)For those who have not received blood transfusions, blood products or blood cytokines such as granulocyte colony-stimulating factor (G-CSF) within 14 days of the first dose, blood routine: neutrophil count ≥2.0×109/L, platelet count ≥100×109 /L, white blood cell count ≥4.0×109/L, hemoglobin concentration ≥8.0g/dL. 2)Blood biochemistry: liver function: aspartate aminotransferase and alanine aminotransferase ≤1.5 times the upper limit of normal (ULN), total bilirubin ≤ULN. kidney function: creatinine ≤1.5×ULN.
5. Baseline left ventricular ejection fraction determined by echocardiography ≥50%, normal or abnormal 12-lead electrocardiogram without clinical significance, QTc interval <450ms (men) or <470ms (women), and no symptoms or signs of heart failure.
6. The functions of major organs (heart, lung, liver, kidney, bone marrow, gastrointestinal) are basically normal or abnormal without clinical significance, and acute toxicity caused by previous treatment is relieved to ≤ grade 1 (except for hair loss).
7. If the subject has been previously treated with surgery, chemotherapy, immunotherapy, biologic therapy, targeted therapy, anti-tumor traditional Chinese medicine, or small molecule targeted drug, the first dose should be given at an interval of 4 weeks or more than 5 half-lives (whichever is shorter)；If the chemotherapeutic agent is mitomycin or nitrosourea, the first dose needs to be given more than 6 weeks apart.
8. The first dose was more than 6 weeks after the last radiotherapy (except palliative radiotherapy for local pain control), and there was no previous whole-pelvic radiotherapy (radiotherapy ≤30% of the bone marrow area).
9. With the consent of the individual and an informed consent form signed by the individual or his legal representative.
10. The subject can communicate well with the researcher and complete the research in accordance with the research regulations.

Exclusion criteria:

1. Those who have received cabazitaxel in the past.
2. Those who are severely allergic to cabazitaxel, human albumin, or alcohol.
3. Currently receiving other anti-tumor therapys.
4. Patients receiving systemic therapy with glucocorticoids (>10 mg/d prednisone or equivalent dose of steroids) or other immunosuppressants within 14 days before the first dose. In the absence of active autoimmune disease, inhaled or topical glucocorticoids can be used, and hormone replacement therapy doses ≤10 mg/d prednisone equivalent are allowed.
5. Those who need to use strong inhibitors or inducers of CYP3A4 within 14 days of the first dose and during the study.
6. Those with clinically significant mental or central nervous system diseases.
7. Those with active brain metastasis.
8. Those with two or more malignant tumors (except cured non-melanoma skin cancer, cervical cancer, thyroid cancer and gastrointestinal intramucosal cancer)
9. Subjects who have received 2 or more prior treatments with mitomycin or nitrosoureas, or subjects who have received prior intensive therapy with autologous stem cell transplantation.
10. Those with serious medical diseases:1)Existence of clinically important cardiovascular and cerebrovascular diseases, including: severe or uncontrollable heart disease that requires treatment, congestive heart failure rated ≥ grade 3 by the New York Heart Association (NYHA), and unstable angina that cannot be controlled by drugs. A history of myocardial infarction within 6 months before enrollment, and severe arrhythmia requiring drug treatment (except for atrial fibrillation or paroxysmal supraventricular tachycardia). 2)Those with indwelling cardiac stent within 6 months.3)Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg), diabetes, pleural effusion, pericardial effusion, and ascites. 4)Uncontrolled peptic ulcer, or other uncontrolled thromboembolic event. 5)Patients with interstitial lung disease, pulmonary fibrosis, or a history of pneumonia who require steroid treatment.
11. People who are infected with HIV, HBV [those who are positive for hepatitis B surface antigen (HBsAg) and whose HBV-DNA is higher than 1000IU/mL], HCV ( those who are HCV-Ab positive and whose HCVRNA detection copy number is higher than normal upper limit)and Treponema pallidum.
12. Those with a history of drug abuse.
13. Women who are pregnant or lactating. female patients of childbearing potential who have a positive pregnancy test within 7 days before the first dose. any male and female patients of childbearing potential do not consent to the use of a medically recognized effective method of contraception throughout the trial and for 3 months after final trial drug administration.
14. Those who have participated in other drug clinical trials within 28 days before the first dose.
15. Those who have been vaccinated within 30 days before the first dose or vaccinated during the study period (except for inactivated vaccines).
16. Other circumstances in which the researcher deems it inappropriate to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluating the tolerability of BH002 in Chinese patients with advanced solid tumors. | 21 days after first dose
  dose-limiting toxicity [DLT]
Evaluating the tolerability of BH002 in Chinese patients with advanced solid tumors. | 21 days after first dose
  maximum tolerated dose [MTD]
Obtain the pharmacokinetic characteristics of BH002 in Chinese patients with advanced solid tumors. | 216 hours after first dose
  Maximum Plasma Concentration [Cmax], etc,

SECONDARY OUTCOMES:
To evaluate the safety of BH002 in Chinese patients with advanced solid tumors. | From first dose to 30 days after last dose
  Rates and severity of adverse events.
Evaluating the preliminary anti-tumor activity of BH002 in Chinese patients with advanced solid tumors | From first dose to 30 days after last dose
  Preliminary observation of the therapeutic effect of the drug.
Determination of recommended phase Ⅱ dose (RP2D) | 21 days after first dose
  Explore clinically applicable doses and dosage regimens in the next phase.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, PI, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No